CLINICAL TRIAL: NCT04292925
Title: Participation and Executive Functions in Adults Following Traumatic Brain Injury During Suba-Acute Inpatient Rehabilitation
Brief Title: Participation and Executive Functions in Adults Following Traumatic Brain Injury In Sub-Acute Inpatient Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Rotem Eliav, Occupational therapist, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0028-18-LOE
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
Keywords: Executive functions; cognitive; sub-acute; rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Intervention with the new treatment protocol will include 18 treatment sessions of 45 minutes, between three to five times a week depending on the participant's state, over a period of four to six weeks.
  Interventions: Other: New treatment protocol
- Control group (Active Comparator): Intervention with conventional therapy will include 18 treatment sessions of 45 minutes, between three to five times a week depending on the participant's state, over a period of four to six weeks.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: New treatment protocol — The new treatment protocol focuses on training of executive processes using remedial strategies and on promoting the use of meta-cognitive strategies. Goal directed activities are used to improve the underlying cognitive process and transfer of the learned skill to everyday function will be encouraged.
  Arms: Experimental Group
Other: Conventional therapy — conventional therapy
  Arms: Control group

SUMMARY:
Aim: To examine the feasibility of a new treatment protocol in improving executive function deficits and participation in daily activities of adults with TBI at discharge and one month post-discharge.

A double-blind (assessors) randomized control trial (RCT) with two groups, experimental and control.

This study will include 40 adults hospitalized in the inpatient Head Trauma unit.

Potential patients will be approached by occupational therapists working in the inpatient Head Trauma rehabilitation unit and be invited to participate in the study. If they agree, they will be asked to sign an informed consent form. Then they will undergo a screening assessment. Participants who are found eligible will be then administered a cognitive assessment battery. Then they will be randomly allocated to either the experimental (new treatment protocol) or the control (conventional therapy) group. In both groups, the intervention will include 18 treatment sessions of 45 minutes, between three to five times a week depending on the participant's state, over a period of four to six weeks. Following the intervention, participants will undergo the assessment again. Participation questionnaires will be administered by telephone one month post-discharge.

DETAILED DESCRIPTION:
A double-blind randomized control trial (RCT) with two groups, experimental and control.

This study will include 40 adults hospitalized in the inpatient Head Trauma unit.

Potential patients will be approached by occupational therapists working in the inpatient Head Trauma rehabilitation unit and be invited to participate in the study. If they agree, they will be asked to sign an informed consent form. Then they will undergo a screening assessment. Participants who are found eligible will be then administered a cognitive assessment battery. Then they will be randomly allocated to either the experimental (new treatment protocol) or the control (conventional therapy) group. In both groups, the intervention will include 18 treatment sessions of 45 minutes, between three to five times a week depending on the participant's state, over a period of four to six weeks. Following the intervention, participants will undergo the assessment again. Participation questionnaires will be administered by telephone one-month post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe TBI as diagnosed by a physician and confirmed by imaging
* age 18-60
* able to understand instructions of assessment tools as will be determined by their Occupational Therapist
* basic cognitive abilities preserved as will be determined by three subtests of the Loewenstein Occupational Therapy Cognitive Assessment: orientation (score: 6/8 or above), visual perception (score: 3/4 or above) and spatial perception (score: 2/4 or above)
* at least one functional upper extremity as will be determined by their Occupational Therapist
* intact or corrected vision.
* a score of 1 or above in the The Multiple Errands Test - the hospital version (MET-HV).

Exclusion Criteria:

* epilepsy
* history of drug use
* other psychiatric or neurologic disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The Multiple Errands Test - the hospital version (MET-HV) | 30 minutes
  A performance-based assessment which was design to assess the effect of EF deficits on everyday functioning.

SECONDARY OUTCOMES:
Cognitive Self Efficacy Questionnaire II (CSEQ) | 15 minutes
  The CSEQ is a questionnaire designed to assess a person's beliefs regarding their ability to recognize, monitor and manage cognitive symptoms and everyday challenging cognitive activities.
Self-Perceptions in Rehabilitation Questionnaire (SPIRQ) | 15 minutes
  The SPIRQ is a 20 items questionnaire designed to measure clients' self-perceptions of injury, perceived benefits of rehabilitation, and emotional reactions throughout inpatient or outpatient rehabilitation.
Mayo-Portland Adaptability Inventory - 4 (MPAI-4) | 15 minutes
  The MPAI is designed to assist in the clinical evaluation of people during post acute period following traumatic brain injury, to assist in the evaluation of rehabilitation programs and to better understand the long-term outcomes of traumatic brain injury.
Quality of Life After Brain Injury (QOLIBRI) | 15 minute
  Is a questionnaire designed to assess quality of life following traumatic brain injury. The QOLIBRI instrument consists of 37 items in four satisfaction scales, ''Cognition'' (7 items), ''Self'' (7 items), ''Daily Life and Autonomy'' (7 items), and ''Social Relationships'' (6 items), and two bothered scales, ''Emotions'' (5 items) and ''Physical Problems'' (5 items).
WebNeuro neurocognitive assessment battery | 30 minutes
  A web-based computerized battery of neurocognitive functioning.

OTHER OUTCOMES:
Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | 30 minutes
  The LOTCA was designed to give a preliminary cognitive profile for patients with an acquired head injury
Functional Independence Measure (FIM) | 15 minutes
  The FIM instrument is designed to assess functional independence. The FIM consists of 18 items which are divided into six subscales (self-care, sphincter control, transfers, locomotion, communication, and social cognition). Each of the 18 items have a maximum score of 7 (complete independence) and a minimum score of 1 (complete dependence), thus possible scores range from 18 to 126 (Donaghy & Wass, 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Rotem Eliav, Principal Investigator — Loewenstein Rehabilitation Hospital
Locations (1):
- Loewenstein Rehabilitation Hospital, Raanana, Israel

REFERENCES:
- [Derived] Eliav R, Nadler Tzadok Y, Segal-Rotenberg S, Kizony R. Efficacy of Intervention of Participation and Executive Functions (I-PEX) for Adults Following Traumatic Brain Injury: A Preliminary Pilot Randomized Controlled Trial. Neurorehabil Neural Repair. 2024 Apr;38(4):279-290. doi: 10.1177/15459683241231529. Epub 2024 Feb 20. PMID 38375580